CLINICAL TRIAL: NCT00961285
Title: High Resolution Genome Wide-Copy Number Profiling and Pharmacogenomic Analysis in Acute Lymphoblastic Leukemia by Single Nucleotide Polymorphism (SNP) Arrays
Brief Title: Genotyping Analysis of Acute Lymphoblastic Leukemia
Acronym: GALL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Giovanni Martinelli, Institute of Hematology "L. & A. Seragnoli" - University of Bologna
Other Study IDs: GENOTYPING ANALYSIS OF ALL
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2009-08

CONDITIONS: Acute Lymphoblastic Leukemia; Adult
Keywords: pharmacogenomics; genotyping
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — extracted DNA or cryopreserved cells in Guanidine isothiocyanate or fresh peripheral blood (10 ml) and/or bone marrow samples (at least 2 ml) in EDTA.
Oversight: Data Monitoring Committee: No

SUMMARY:
Identification of alterations potentially involved in the complex mechanisms of leukemogenesis and at the identification and validation of novel biological factors which may serve as predictors of drug-response and drug-resistance or which may be suitable for targeted therapy.

DETAILED DESCRIPTION:
The investigators will use several approach to identify common genetic variations: single-nucleotide polymorphisms (SNPs), genomic insertions and deletions, and genetic copy number variations (CNVs), interchromosomal translocations, loss of heterozygosity (LOH), and uniparental disomy (UPD), Epigenetic changes, such as silencing of gene expression via DNA hypermethylation, that can also influence drug effects, and aberrant methylation of CpG islands is a common feature of cancer cells. Over the years, methods of cytogenetic analysis evolved and became part of routine laboratory testing, providing valuable diagnostic and prognostic information in hematologic disorders. The recently developed single nucleotide polymorphism (SNP) arrays offer the ability to define simultaneously the copy number changes and loss of heterozygosity (LOH) events occurring in a tumor, at high resolution and throughout the genome. In addition to information on copy number changes, SNP arrays allow us to investigate the impact of a high number of SNPs on drug response and toxicity This molecular integrated approach will lead to the identification of alterations potentially involved in the complex mechanisms of leukemogenesis and at the identification and validation of novel biological factors which may serve as predictors of drug-response and drug-resistance or which may be suitable for targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute Lymphoblastic Leukemia of any subtype OR Lymphoid blast crisis Chronic Myeloid Leukemia
* Age > 18 years
* Available data set of clinical data for review (demographics including ethnicity, stage of disease, concise treatment history, cytogenetic reports, and molecular results if available as routinely performed during diagnosis procedures)

Inclusion Criteria:

* No written informed consent
* No DNA samples available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult ALL patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To provide high resolution molecular karyotyping analysis by single nucleotide polymorphism array (SNP 6.0, Affymetrix) of adult patients with diagnosis of acute lymphoblastic leukemia (ALL), newly enrolled in clinical trials | December 2011

SECONDARY OUTCOMES:
To study by pharmacogenomic analysis based on SNPs profile, and predict the individual susceptibility (i.e. efficacy and toxicity) to therapeutic treatment and disease development | December 2011
To identify useful biomarkers for disease outcome and disease progression | December 2011
To identify useful biomarkers related to drug exposure or to response to potential toxic drugs | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, prof., Principal Investigator — University of Bologna
Locations (1):
- Institute of Hematology "L. & A. Seragnoli", Bologna, Italy